CLINICAL TRIAL: NCT03210376
Title: The Effect of Deep Neuromuscular Blockade With Sugammadex Reversal on Shoulder Pain of Elderly Patients Undergoing Robotic Surgery: A Single-Center Double-Blinded Randomized Controlled Trial
Brief Title: Neuromuscular Blockade on Shoulder Pain of Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-0046; NCI-2018-01176 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-06-29; First posted 2017-07-06 (Actual); Results first posted 2019-10-07 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Malignant Neoplasms of Digestive Organs; Malignant Neoplasms of Female Genital Organs; Malignant Neoplasms of Male Genital Organs; Malignant Neoplasms of Urinary Tract
Keywords: Malignant neoplasms of digestive organs; Malignant neoplasms of female genital organs; Malignant neoplasms of male genital organs; Malignant neoplasms of urinary tract; Neuromuscular blockade; NMB; Sugammadex; Neostigmine; Pain Assessment; Survey
MeSH Terms: conditions — Urologic Neoplasms | interventions — Sugammadex; Neostigmine; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep Neuromuscular Blockade (NMB) + Sugammadex (Experimental): Deep Neuromuscular Blockade (NMB) given during surgery.
  Sugammadex intravenously as a single bolus injection after surgery.
  Pain assessment done at about 15, 45, and 90 minutes after surgery.
  Interventions: Drug: Deep Neuromuscular Blockade (NMB); Drug: Sugammadex; Behavioral: Pain Assessment
- Moderate Neuromuscular Blockade (NMB) + Neostigmine (Experimental): Moderate Neuromuscular Blockade (NMB) given during surgery.
  Neostigmine intravenously slowly over a period of at least 1 minute after surgery.
  Pain assessment done at about 15, 45, and 90 minutes after surgery.
  Interventions: Drug: Moderate Neuromuscular Blockade (NMB); Drug: Neostigmine; Behavioral: Pain Assessment

INTERVENTIONS:
Drug: Deep Neuromuscular Blockade (NMB) — Deep Neuromuscular Blockade (NMB) given during surgery.
  Arms: Deep Neuromuscular Blockade (NMB) + Sugammadex
Drug: Moderate Neuromuscular Blockade (NMB) — Moderate Neuromuscular Blockade (NMB) given during surgery.
  Arms: Moderate Neuromuscular Blockade (NMB) + Neostigmine
Drug: Sugammadex — 4 mg/Kg, intravenously as a single bolus injection after surgery.
  Arms: Deep Neuromuscular Blockade (NMB) + Sugammadex
Drug: Neostigmine — 70 mcg/Kg up to a total of 5 mg, intravenously slowly over a period of at least 1 minute after surgery.
  Arms: Moderate Neuromuscular Blockade (NMB) + Neostigmine
Behavioral: Pain Assessment — Pain assessment done at about 15, 45, and 90 minutes after surgery.
  Other Names: Survey

SUMMARY:
Insufflation pressure (IP) is the creation of a pressure barrier of air/gas within the abdomen to allow the surgeon more space to work during abdominal surgery. Shoulder pain is a common complaint from patients who have had abdominal surgery and the pain is thought to be related to the use of IP.

In addition to anesthesia (which keeps you asleep during surgery), the current standard practice is to block the nerve-muscle junction with a type of drug called neuromuscular blockade (NMB) which paralyzes the abdominal muscles. This means that a lower level of insufflation pressure is needed by the surgeon.

To reverse the effects of NMB after surgery, a drug called neostigmine is given.

The goal of this clinical research study is to compare the use of standard-of-care moderate NMB and neostigmine to the use of deep NMB and a drug called Sugammadex when given to elderly patients (patients who are 65 years of age or older) who are scheduled to have robotic abdominal surgery. "Deep" and "moderate" in this study refers to the dose or strength of the NMB given.

This is an investigational study. Sugammadex and neostigmine are FDA approved and commercially available for the reversal of NMB. It is considered investigational to compare Sugammadex and neostigmine to learn if the use of one or the other in elderly patients can reduce the level of shoulder pain after surgery.

Up to 100 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups before your surgery. This is done because no one knows if one group is better, the same, or worse than the other.

* In Group 1, you will receive deep NMB and Sugammadex.
* In Group 2, you will receive moderate NMB and neostigmine.

Neither you nor the surgeon or surgical staff will know to which group you have been assigned. The surgeon will not know which group you are in because researchers want to learn how much, if at all, the surgeon needs to adjust the insufflation pressure during surgery. However, if needed for your safety, the surgeon will be able to find out which group you are in.

For your safety, the anesthesiologist will know to which group you have been assigned.

Surgery and Study Drug Administration:

After you have been assigned to a study group, you will have your surgery as scheduled. You will sign a separate consent form for surgery which describes the procedure and its risks in more detail. You will also sign a separate consent form to receive anesthesia.

Before your surgery, blood (about 2 teaspoons) will be drawn for biomarker testing. Biomarkers are found in the blood/tissue and may be related to the status of the disease and/or your reaction to the study drug(s).

During the surgery, the insufflation pressure that is being used, including any changes that are made to the pressure, will be recorded. After the surgery has been completed, you will receive either Sugammadex or neostigmine by vein until the effects of the NMB have been reversed.

You will recover after surgery in the post-anesthesia care unit (PACU). At about 15, 45, and 90 minutes after your surgery, a PACU nurse will ask you about any shoulder pain you are feeling and if so, how intense the pain is. Information about how long you stay in the hospital after surgery and if you have any side effects after surgery (such as nausea/vomiting or shoulder pain) will also be collected from your medical record.

Follow-Up:

After 30 days after you leave the hospital, you will be called by a member of the study staff to ask how you are doing and if you have had any additional hospitalizations since leaving the hospital. This phone call should last about 5-10 minutes.

Length of Study Participation:

Your participation in this study will be over after completing the 30-day follow up phone call.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 65 years of age or older
2. Patients having robotic prostatectomy
3. Written informed consent

Exclusion Criteria:

1. Patient with known hypersensitivity to Rocuronium, Sugammadex or its components
2. Patients with severe renal insufficiency, defined and confirmed by an estimated creatinine clearance equal or lower than 30 mL/min, per institutional laboratory.
3. Patients with history of severe liver disease, defined as and confirmed by elevated ALT and AST greater than 1.5 times the Upper Limit of Normal along with Albumin less than 3 OR INR 1.5 or greater per institutional laboratory.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2020-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendell H. Williams III, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Williams WH 3rd, Cata JP, Lasala JD, Navai N, Feng L, Gottumukkala V. Effect of reversal of deep neuromuscular block with sugammadex or moderate block by neostigmine on shoulder pain in elderly patients undergoing robotic prostatectomy. Br J Anaesth. 2020 Feb;124(2):164-172. doi: 10.1016/j.bja.2019.09.043. Epub 2019 Nov 26. PMID 31780139
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were identified when scheduled for Robotic Prostatectomy. Eligible subjects were approached before scheduled surgery to obtain Informed Consent. Patients were recruited from November, 2017 through July, 2018.
Groups:
- Deep Neuromuscular Blockade (NMB) + Sugammadex: The patients will be started on a continuous Rocuronium intravenous infusion following intubation. Insert recommendations and Institutional Standards will be used for Rocuronium. For the DNMB group, the rate will be adjusted and boluses given to maintain 1-2 post tetanic responses during the pneumoperitoneum. NMB will be reversed with Sugammadex 4 mg/Kg, intravenously as a single bolus injection, at the end of the surgery.
- Moderate Neuromuscular Blockade (NMB) + Neostigmine: The patients will be started on a continuous Rocuronium intravenous infusion following intubation. Insert recommendations and Institutional Standards will be used for Rocuronium. For the MNMB group, the Rocuronium infusion rate will be adjusted to maintain 1-2 TOF responses and will be reversed with Neostigmine 70 mcg/Kg up to a total of 5 mg, intravenously slowly over a period of at least 1 minute, at the end of surgery.
Period: Overall Study
Arm/Group | Deep Neuromuscular Blockade (NMB) + Sugammadex | Moderate Neuromuscular Blockade (NMB) + Neostigmine
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Blockade (NMB) + Sugammadex | Moderate Neuromuscular Blockade (NMB) + Neostigmine | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 44 | 43 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.12 (3.6289) | 69.26 (3.6073) | 69.19 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 50 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 44 | 42 | 86
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 40 | 39 | 79
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.044 (4.8) | 28.662 (3.9567) | 28.85 (4.38)
Adjuvant or Immunotherapy [Count of Participants; unit: Participants] | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Reported Shoulder Pain
Description: Visual Analog Scale (VAS) pain score (0-10) for shoulder pain recorded, where 0 means no pain and 10 means the worst pain ever experienced . Percentage of participants who experienced should pain.
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Deep Neuromuscular Blockade (NMB) + Sugammadex | Moderate Neuromuscular Blockade (NMB) + Neostigmine
Number analyzed (Participants) | 50 | 50
percentage of participants | 12 | 10

2. Secondary Outcome: Cumulative Intraoperative Insufflation Pressure
Description: Intra-abdominal insufflation time and pressure directed by the surgeon and recorded continuously by the clinical coordinator until the time of desufflation.
Time Frame: Day 0 - IntraOperative-From beginning of pneumoperitoneum to desufflation (an average of 166 minutes)
Measure: Median (Full Range); unit: mmHg
Arm/Group | Deep Neuromuscular Blockade (NMB) + Sugammadex | Moderate Neuromuscular Blockade (NMB) + Neostigmine
Number analyzed (Participants) | 50 | 50
mmHg | 1995 [1104 to 3550] | 1581 [870 to 3555]

3. Secondary Outcome: Percentage of Muscle Response Using Train-of-Four (TOF) in Post-Anesthesia Care Unit (PACU) to Measure Residual Muscle Relaxation
Description: The patients will be started on a continuous Rocuronium intravenous infusion following intubation. Insert recommendations and Institutional Standards will be used for Rocuronium. For the DNMB group, the rate will be adjusted and boluses given to maintain 1-2 post tetanic responses during the pneumoperitoneum. NMB will be reversed with Sugammadex 4 mg/Kg, intravenously as a single bolus injection, at the end of the surgery. Percentage of measured contraction strength of the fourth stimulus compared to the first stimulus.
Time Frame: Day 0 - Arrival time at PACU, an average of 3 minutes
Measure: Median (Full Range); unit: Percentage of measured contraction
Arm/Group | Deep Neuromuscular Blockade (NMB) + Sugammadex | Moderate Neuromuscular Blockade (NMB) + Neostigmine
Number analyzed (Participants) | 50 | 50
Percentage of measured contraction | 110 [70 to 174] | 100 [50 to 155]

4. Secondary Outcome: Readiness to Discharge From the Post-Anesthesia Care Unit (PACU)
Description: Determined by the Dansk Selskab for Anæstesiologi og Intensiv Medicin(DASAIM)discharge criteria.Pts considered ready to discharge when the sum of all categories is<4 and no single category has a score of >1.Sedation.0:Patient is fully awake.1: Patient is asleep,aroused by verbal stimulation.2:Patient is asleep, aroused by physical stimulation.3:Patient is asleep,cannot be aroused.Respiratory Rate.0:Respiratory rate>10. 1: Snoring,10< RR<30. 2:R<10 or RR>30/min.3:Periods of apnea or obstructive patterns.Oxygen Saturation.0:SpO2 ≥ 94%.1:90%≤SpO2<94%. 2:85%≤ SpO2 < 90%.3:SpO2 < 85%. Systolic Blood Pressure. 0:SBP ≥ 100mmHg.1:90mmHg≤SBP< 100mmHg.2:80mmHg≤SBP< 90mmHg or SBP>220mmHg.3:SBP<80mmHg.Heart Rate.0:50<HR≤100.1:100<HR≤120.2:40<HR≤ 50 or 120<HR≤130.3:HR<40 or HR>130.Pain at rest.0:No pain 1:Light pain.2:Moderate pain.3:Severe pain.Nausea.0:No nausea or vomiting.1:Light nausea or vomiting without previous nausea. 2:Moderate nausea and/or vomiting.3:Severe nausea and/or vomiting.
Time Frame: Assessed at 15, 45, 90 minutes during PACU stay.
Measure: Median (Standard Deviation); unit: Score on a scale
Arm/Group | Deep Neuromuscular Blockade (NMB) + Sugammadex | Moderate Neuromuscular Blockade (NMB) + Neostigmine
Number analyzed (Participants) | 50 | 50
Score on a scale
  DASAIM at 15 min | 2.92 (1.6393) | 3.16 (1.6946)
  DASAIM at 45 min | 2.82 (1.6744) | 2.86 (1.6904)
  DASAIM at 90 min | 2.12 (1.599) | 1.8 (1.4286)

5. Secondary Outcome: Percentage of Participants With Nausea and/or Vomiting in PACU
Description: Degree of Post-Operative Nausea determined per Visual Analog Scale per nurse in Post-Anesthesia Care Unit (PACU).
Time Frame: Day 0 - PACU stay, an average of 120 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Deep Neuromuscular Blockade (NMB) + Sugammadex | Moderate Neuromuscular Blockade (NMB) + Neostigmine
Number analyzed (Participants) | 50 | 50
percentage of participants
  Nausea | 7 | 6
  Vomiting | 1 | 0

6. Secondary Outcome: Surgical Exposure Grading
Time Frame: Day 0 - IntraOperative, from incision time to closing time(average 190 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Deep Neuromuscular Blockade (NMB) + Sugammadex | Moderate Neuromuscular Blockade (NMB) + Neostigmine
Number analyzed (Participants) | 50 | 50
Participants
  Optimal | 25 | 33
  Good | 19 | 8
  Acceptable | 5 | 8
  Poor | 1 | 1

7. Secondary Outcome: Length of Hospital Stay
Time Frame: length of hospital stay(average of 3 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Deep Neuromuscular Blockade (NMB) + Sugammadex | Moderate Neuromuscular Blockade (NMB) + Neostigmine
Number analyzed (Participants) | 50 | 50
days | 2.2323 (2.0859) | 1.8623 (1.0545)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Deep Neuromuscular Blockade (NMB) + Sugammadex | Moderate Neuromuscular Blockade (NMB) + Neostigmine
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50 | 2/50
Other Adverse Events (participants affected / at risk) | 13/50 | 15/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deep Neuromuscular Blockade (NMB) + Sugammadex (N=50) | Moderate Neuromuscular Blockade (NMB) + Neostigmine (N=50)
Chest Pain (Cardiac disorders) | 1 | 0
Incarcerated Inguinal Hernia (Musculoskeletal and connective tissue disorders) | 1 | 0
Partial Small Bowel Obstruction (Gastrointestinal disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1
Anastomosis Leak (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deep Neuromuscular Blockade (NMB) + Sugammadex (N=50) | Moderate Neuromuscular Blockade (NMB) + Neostigmine (N=50)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Chest Pain (Cardiac disorders) | 1 | 0
Fever (Immune system disorders) | 1 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Postoperative Ileus (Gastrointestinal disorders) | 4 | 1
Urinary Tract Infection (Renal and urinary disorders) | 4 | 3
Low O2 Sat (Vascular disorders) | 0 | 1
Infected Incision (Skin and subcutaneous tissue disorders) | 0 | 1
Uncontrolled Hypertension (Vascular disorders) | 0 | 1
Restlessness Legs (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT03210376/Prot_SAP_000.pdf